CLINICAL TRIAL: NCT00737529
Title: A Phase 2, Multicenter, Single-Arm, Open-Label Study To Determine The Efficacy And Safety Of Single-Agent Lenalidomide (Revlimid®) In Patients With Mantel Cell NHL Who Have Relapsed Or Progressed After Treatment With Bortezomib Or Are Refractory To Bortezomib
Brief Title: A Study to Determine the Efficacy and Safety of Lenalidomide in Patients With Mantle Cell NHL Who Have Relapsed or Progressed After Treatment With Bortezomib or Are Refractory to Bortezomib. The "EMERGE" Trial
Acronym: EMERGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MCL-001
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; CC-5013; Revlimid; Lenalidomide
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Single agent Lenalidomide
  Lenalidomide: 10mg or 25 mg oral capsules on days 1 to 21 of each 28 day cycle and dependent on renal function; Participants with normal renal function (defined as Creatinine Clearance(CrCl)) of ≥ 60 mL/min in this study) received 25 mg of lenalidomide daily, and those with moderate renal insufficiency (CrCl) ≥ 30 mL/min but < 60 mL/min) were started at a 10-mg dose. Participants could continue to receive treatment until disease progression, development of unacceptable AEs, or voluntary withdrawal.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — 25mg oral capsules continuous days 1-21 each of a 28 day cycle
  Other Names: Revlimid

SUMMARY:
To evaluate the safety and efficacy of Lenalidomide (Revlimid (R)) in subjects with mantle cell lymphoma who have relapsed, progressed or are refractory to bortezomib.

DETAILED DESCRIPTION:
Follow up phase will continue until either 100% of the patients have died, are lost to follow up or have withdrawn consent or a maximum of 4 years from the last patient enrolled, whichever comes first. All other efficacy and safety endpoints will be updated at this time. In the unlikely event that the study will be closed and patients are still responding to treatment at this time, Celgene will discuss with the treating physicians options to provide further treatment to the patient after study closure in line with local regulation.

Follow up for second primary malignancies and OS will continue until 100% of the patients have died, are lost to follow up, have withdrawn consent, or a maximum of 5 years from the last patient enrolled, whichever comes first.

10 October 2017: In regard to the last subject last visit date/study completion date, the prolongation of timelines is due to the bridging of a treatment gap for a patient responding to study medication until non-study medication is available.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven mantle cell lymphoma
* Patients must have documents relapsed, refractory or PD after treatment with bortezomib
* Must have measureable disease on cross sectional imaging by CT
* Eastern Cooperative Oncology Group (ECOG) performance score 0,1 or 2
* Willing to follow pregnancy precautions

Exclusion Criteria:

* Any of the following laboratory abnormalities

  * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L)
  * Platelet count < 60,000/mm3 (60 x 109/L)
  * Serum aspartate transaminase/Serum glutamic oxaloacetic transaminase(AST/SGOT) or alanine transaminase/Serum glutamic pyruvic transaminase (ALT/SGPT) > 3.0 x upper limit of normal (ULN), except in patients with documented liver involvement by lymphoma.
  * Serum total bilirubin > 1.5 x ULN, except in cases of Gilbert's Syndrome and documented liver involvement by lymphoma.
  * Calculated creatinine clearance (Cockcroft-Gault formula) of < 30 mL /min
  * Patients who are candidates for high dose chemotherapy/allogeneic stem cell transplant are not eligible
  * History of active central nervous system (CNS) lymphoma within the previous 3 months
  * Subjects not willing or unable to take deep vein thrombosis (DVT) prophylaxis
  * Prior history of malignancies, other than MCL, unless the patient has been free of the disease for ≥ 3 years
  * Positive Human immunodeficiency virus (HIV) or active Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-12-22 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Director — Celgene Corporation
Locations (70):
- United States (31):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCSD Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Tower Cancer Research Foundation, Los Angeles, California
  - Boca Raton Community Hospital, Inc., Research Dept., Boca Raton, Florida
  - Pasco Hernando Oncology Associates, PA, Brooksville, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - MD Anderson Cancer Center, Orlando Regional Healthcare, Orlando, Florida
  - Lake County Oncology and Hematology, The Villages, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center - Smith, Maywood, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Alvin and Lois Lapidus Cancer Institute Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU School of Medicine, New York, New York
  - University of Rochester Cancer Center, James P. Wilmot Cancer Center, Rochester, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Hillman Cancer Institute at UPMC, Pittsburgh, Pennsylvania
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - University of Virginia Cancer Center Clinical Trials Office, Charlottesville, Virginia
- Austria (3):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (3):
  - AZ Sint-Jan AV Brugge, Bruges
  - UZ Gent, Ghent
  - Universitair Ziekenhuis Leuven, Campus Gasthuisberg, Leuven
- Colombia (2):
  - Hospital Universitario San Ignacio, Bogotá
  - Oncologos del occidente S.A., Pereira
- France (9):
  - Hopital Sud, CHU d'Amiens, Amiens
  - Institut Bergonie, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Hopital Emile Muller, Mulhouse
  - Hopital Cochin, Paris
  - Institut Curie, Paris
  - Hopital Robert Debre, Reims
  - Institut de Cancerologie de la Loire, Saint Jean Priest En Jarez
  - Hopital Hautepierre, Strasbourg
- University Hospital Wuerzburg, Würzburg, Germany
- Hungary (4):
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - University of Debrecen, DEOEC, Institute of Internal Medicine, Debrecen
  - Petz Aladar Megyei Oktato Korhaz,II. Belgyogyaszat, Győr
  - Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petch Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Universita Federico II di Napoli Nuovo Policlinico, Napoli
  - Ospedale Civile dello Spirito Santo, Pescara
  - Universita Cattololica del Sacro Cuore, Roma
- Centro De Cancer, Hospital Espanol Auxilio De Puerto Rico, San Juan, Puerto Rico
- Singapore General Hospital, Singapore, Singapore
- Spain (4):
  - Hospital General De Elche, Alicante
  - Duran i Reynals Institut Catala d'Oncologia, L'Hospitalet de Llobregat
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario La Fe, Valencia
- Turkey (Türkiye) (3):
  - Gazi Universitesi, Besevler Ankara
  - Istanbul Universitesi Istanbul, Istanbul
  - Ankara Universitesi Tip Fakultesi, Sihhiye Ankara
- Royal Cornwall Hospitals Trust, Truro, United Kingdom

REFERENCES:
- [Background] Goy A, Sinha R, Williams ME, Kalayoglu Besisik S, Drach J, Ramchandren R, Zhang L, Cicero S, Fu T, Witzig TE. Single-agent lenalidomide in patients with mantle-cell lymphoma who relapsed or progressed after or were refractory to bortezomib: phase II MCL-001 (EMERGE) study. J Clin Oncol. 2013 Oct 10;31(29):3688-95. doi: 10.1200/JCO.2013.49.2835. Epub 2013 Sep 3. PMID 24002500
- [Result] Goy A, Kalayoglu Besisik S, Drach J, Ramchandren R, Robertson MJ, Avivi I, Rowe JM, Herbrecht R, Van Hoof A, Zhang L, Cicero S, Fu T, Witzig T. Longer-term follow-up and outcome by tumour cell proliferation rate (Ki-67) in patients with relapsed/refractory mantle cell lymphoma treated with lenalidomide on MCL-001(EMERGE) pivotal trial. Br J Haematol. 2015 Aug;170(4):496-503. doi: 10.1111/bjh.13456. Epub 2015 Apr 28. PMID 25921098
- [Result] Witzig TE, Luigi Zinzani P, Habermann TM, Tuscano JM, Drach J, Ramchandren R, Kalayoglu Besisik S, Takeshita K, Casadebaig Bravo ML, Zhang L, Fu T, Goy A. Long-term analysis of phase II studies of single-agent lenalidomide in relapsed/refractory mantle cell lymphoma. Am J Hematol. 2017 Oct;92(10):E575-E583. doi: 10.1002/ajh.24854. Epub 2017 Aug 28. PMID 28699256
- [Derived] San-Miguel JF, Richardson PG, Gunther A, Sezer O, Siegel D, Blade J, LeBlanc R, Sutherland H, Sopala M, Mishra KK, Mu S, Bourquelot PM, Victoria Mateos M, Anderson KC. Phase Ib study of panobinostat and bortezomib in relapsed or relapsed and refractory multiple myeloma. J Clin Oncol. 2013 Oct 10;31(29):3696-703. doi: 10.1200/JCO.2012.46.7068. Epub 2013 Sep 9. PMID 24019544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated at 42 centers in 12 countries: US/ Puerto Rico, France, Israel, Belgium, Spain, Turkey, Austria, Hungary, Italy, Colombia, Germany, and Singapore.
Pre-assignment Details: All participants were required to have local histologic confirmation of Mantle Cell Lymphoma (MCL) for entry into the study.
Groups:
- Lenalidomide: Participants received lenalidomide 10 mg or 25 mg oral capsules on days 1 to 21 of each 28-day cycle and was dependent on renal function; Participants with normal renal function (defined as creatinine clearance (CrCl)) of ≥ 60 mL/min) received 25 mg of lenalidomide by mouth (PO) daily, and those with moderate renal insufficiency (CrCl) ≥ 30 mL/min but < 60 mL/min) were started at a 10 mg daily dose. Participants could continue to receive treatment until disease progression, development of unacceptable adverse events (AEs), or voluntary withdrawal.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 134
Completed | 1 (Completed equals participants ongoing on treatment at the time of the data cut-off of 30 March 2017)
Not Completed | 133
Not completed — Disease Progression | 95
Not completed — Adverse Event | 24
Not completed — Withdrawal by Subject | 5
Not completed — Death | 4
Not completed — Protocol Violation | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are from the participants assesed within the intent to treat population (ITT), which included all enrolled participants who received at least one dose of study drug.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.38)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 49
  ≥ 65 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 128
  Asian | 3
  Black or African American | 1
  Other | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = (Fully Active) | 43
    1 = (Restrictive but ambulatory) | 73
    2 = (Ambulatory but unable to work) | 17
    3 = (Limited self care) | 1
    4 = (Completely Disabled) | 0
Renal function at baseline [Count of Participants; unit: Participants] — Participants with a Creatinine clearance (as calculated by the Cockcroft-Gault formula, utilizing actual body weight or ideal body weight, whichever was less) of ≥ 60 mL/min received a starting dose of 25 mg once daily. Participants with moderate renal insufficiency (ie, CrCl ≥ 30 mL/min but < 60 mL/min) received a starting dose of 10 mg lenalidomide once daily.
  Participants
    Normal (CrCl > = 60 mL/min) | 99
    Moderate Renal Insufficiency (CrCl ≥ 30 and < 60mL | 28
    Severe Renal Insufficiency (CrCl < 30 mL/min) | 1
    Missing | 6
Duration of Mantle Cell Lymphoma [Number; unit: years]
  <3 years | 52
  ≥ 3 years | 82
MCL (Ann Arbor) Stage at Diagnosis [Count of Participants; unit: Participants] — Ann Arbor staging is the staging system for lymphomas, both in Hodgkin's lymphoma (previously called Hodgkin's disease) and Non-Hodgkin lymphoma (NHL). Stage I = Involvement of 1 Lymph Node (LN) or extralymphatic region; Stage II = ≥ 2 LN sites on the same side of the diaphragm; Stage III = LN regions on both sides of the diaphragm; may include spleen and 1 extralymphatic organ; Stage IV = involvement of ≥ 1 extralymphatic organs with or without associated LN involvement (diffuse or disseminated).
  Participants
    I | 2
    II | 5
    III | 19
    IV | 105
    Missing | 3
MCL International Prognostic Index (MIPI) Score Group at Enrollment [Count of Participants; unit: Participants] — A prognostic index predictive of the outcome in advanced Mantle Cell Lymphoma
  Participants
    Low | 39
    Intermediate | 51
    High | 39
    Missing | 5
Prior Bone Marrow Assessment [Count of Participants; unit: Participants] — Baseline assessment of bone marrow involvement was not required per protocol; however, bone marrow biopsy and aspirate data previously conducted were collected if available.
  Participants
    Positive | 55
    Negative | 52
    Indeterminate | 8
    Missing | 19
Tumor Burden [Count of Participants; unit: Participants] — Defined as at least one lesion that was ≥ 5 cm in diameter or ≥ 3 lesions that were ≥ 3 cm in diameter by central radiology review.
  Participants
    High = having 1 lesion ≥ 5 cm or 3 lesions ≥ 3cm | 78
    Low = < 5cm lesions | 54
    Missing = unable to characterize | 2
Bulky Disease [Count of Participants; unit: Participants] — Bulky disease is defined as at least one lesion ≥ 7 cm in diameter
  Participants
    Yes | 44
    No | 88
    Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Overall Response According to the Independent Review Committee (IRC)
Description: Overall Response Rate (ORR) was defined as the percentage of participants whose best response was Complete Response, Complete Response unconfirmed or Partial Response. Participants who had discontinued before any response has been observed, or changed to other anti-lymphoma treatments before response had been observed, were considered as non-responders. Tumor Response was assessed by a modification of the International Lymphoma Workshop Response Criteria, IWRC, Cheson, 1999); CR is defined as the disappearance of all clinical and radiographic evidence of disease; CRu is defined as a CR, with a 1) residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters (SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2) indeterminate bone marrow; PR = is defined ≥50% decrease in 6 largest nodes or nodal masses.
Time Frame: From Day 1 of study treatment to progession or early treatment discontinuation; up to data cut-off date of 06 April 2016; median duration of treatment was 94.5 days.
Population: ITT population defined as all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
percentage of participants | 29.9 [22.26 to 38.36]

2. Primary Outcome: Kaplan Meier Estimate of Duration of Response (DoR) According to the Independent Review Committee
Description: Kaplan Meier estimate for the duration of response (DoR) was calculated from the date of the first occurrence of initial response for responders (demonstrating evidence of at least a PR) to the date of first documented disease progression (any new lesion or increase by ≥ 50% of previously involved sites from nadir) or death (without documented progression) for participants who responded; participants who had not progressed (or died) were censored at the last valid assessment.
Time Frame: From Day 1 of study drug to progression or early treatment discontinuation; up to data cut-off date of 06 April 2016; Median duration of treatment was 94.5 days.
Population: Includes participants from the ITT population who achieved a PR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 40
months | 16.64 [10.4219 to 29.8191]

3. Secondary Outcome: Percentage of Participants With a Complete Response (CR) /Complete Response Unconfirmed (CRu) According to the Independent Review Committee
Description: The percentage of participants whose best response was CR or CRu. Participants who had discontinued before CR/CRu was observed, or changed to other anti-lymphoma treatments before a CR/CRu response had been observed, were considered as non-responders. CR is defined as the disappearance of all clinical and radiographic evidence of disease; CRu is defined as a CR, with a 1) residual lymph node mass >1.5 cm that has decreased by 75% in the sum of the product of the diameters (SPD). Individual nodes previously confluent decreased by more than 75% in the SPD compared with original mass; 2) indeterminate bone marrow.
Time Frame: as for outcome 2
Population: The ITT population was defined as all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
percentage of participants | 9.0 [4.71 to 15.12]

4. Secondary Outcome: Kaplan Meier Estimate of Duration of Complete Response (DoCR) (CR+CRu) According to the Independent Review Committee
Description: Kaplan Meier estimates for the duration of CR/CRu was calculated from the date of the first occurrence of CR/CRu to the date of documented disease progression or death (without documented progression) for participants who obtained a CR/CRu; participants who had not progressed (or died) were censored at the last valid assessment.
Time Frame: From Day 1 of study drug to progression or early discontinuation; up to data cut-off date of 06 April 2016; median time in follow-up was 16.34 months
Population: Includes participants from the ITT population who achieved a CRu or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
months | 24.43 [5.063 to NA] — NA indicates the upper limit of DoR of CR+CRu was not estimable at final cut-off date as of 06 April 2016 due to participants remaining on study.

5. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) According to the Independent Review Committee
Description: Kaplan Meier estimates of PFS was defined as the start of study drug therapy to the first observation of disease progression or death due to any cause, whichever comes first. If a participant had not progressed or died, PFS was censored at the time of last adequate assessment when the participant was known not to have progressed. For participants who received other anti-lymphoma therapy with no evidence of progression, PFS was censored at time of last adequate tumor assessment with no evidence of progression prior to the start of new anti-lymphoma treatment.
Time Frame: From Day 1 of study drug to first documented date of disease progression; up to data cut-off date of 06 April 2016; median time in follow-up was 16.34 months
Population: Intent to Treat population defined as all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
months | 4.01 [3.6822 to 7.2329]

6. Secondary Outcome: Kaplan Meier Estimate of Time to Progression (TTP) According to the Independent Review Committee
Description: Kaplan Meier estimate of time to progression was calculated as time from the start of the study drug therapy to the first observation of disease progression. Participants who died without progression were censored at the date of death; otherwise, the censoring rules presented above for PFS applied to the analysis of TTP. Progressive Disease(PD): Appearance of new lesion or increase by ≥50% from previously involved sites from nadir
Time Frame: From Day 1 of study drug to first documented time of progression; up to data cut-off date of 06 April 2016; median time in follow-up was 16.34 months
Population: Intent to Treat population was defined as all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
months | 5.46 [3.7479 to 9.4685]

7. Secondary Outcome: Kaplan-Meier Estimate of Time to Treatment Failure (TTF) According to the Independent Review Committee
Description: Time to treatment failure (TTF) was calculated from the start of study drug therapy to early discontinuation from treatment due to any cause, including disease progression, toxicity, or death and was based on site-reported data.
Time Frame: From Day 1 of study drug to first documented time of treatment failure; up to data cut-off date of 06 April 2016; median duration of treatment was 94.5 days
Population: Intent to Treat population was defined as all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
months | 3.75 [2.3342 to 4.6356]

8. Secondary Outcome: Time to Response (TTR)
Description: Time to Response was defined as the time from first dose of study drug to the date of the first response (having at least a PR) and was calculated only for responding participants.
Time Frame: From Day 1 of study drug to time of first documented PR or better; up to data cut-off date of 06 April 2016; median duration of treatment was 94.5 days
Population: Included participants from the ITT population who achieved a PR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 40
months | 3.5 [1.7 to 15.9]

9. Secondary Outcome: Time to Complete Response (CR+CRu) According to the Independent Review Committee
Description: Time to Complete Response (CR+CRu) was defined as the time from the first dose of study drug to the date of the first occurrence of at least CRu and was calculated only for participants with CR or CRu.
Time Frame: From Day 1 of study drug to first documented CR/CRu or better; up to data cut-off date of 06 April 2016; median duration of treatment was 94.5 days
Population: Included participants from the ITT population who achieved a CRu or better.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
months | 3.9 [1.9 to 13.0]

10. Secondary Outcome: Overall Survival (OS)
Description: Kaplan Meier estimate of overall survival was calculated from the time the first dose of study drug to death from any cause. Participants who had not died were censored at the last date the participant was known to be alive.
Time Frame: From Day 1 of study drug to first documented date of progressive disease or death; up to the final data cut-off date of 30 March 2017; median duration of follow-up for surviving participants was 62.94 months
Population: Intent to Treat population defined as all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
months | 19.50 [13.6767 to 25.5781]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events were assessed using National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 3: according to the following scale: Grade 1 = Mild Adverse Event (AE), Grade 2 = Moderate AE, Grade 3 = Severe and Undesirable AE, Grade 4 = Life-threatening or Disabling AE, and Grade 5 = Death; Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above. after the first dose of study drug and within 28 days after the last dose. A TEAE is defined as any AE occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug.
Time Frame: From the first dose of lenalidomide through 28 days after the last dose during the follow-up phase; median (minimum, maximum) duration of treatment was 94.0 (1.0, 1950 days)
Population: The safety population received at least one dose of lenalidomide was used for all safety analysis. This was identical to the ITT population.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 134
participants
  Any TEAE | 132
  Any TEAE Related to Investigational Product (IP) | 118
  Any TEAE Grade 3-5 AE | 106
  Any TEAE Grade 3 AE | 101
  Any TEAE Grade 4 AE | 57
  Any TEAE Grade 5 AE | 18
  Any Grade 3-5 AE Related to IP | 90
  Any Grade 3 AE Related to IP | 88
  Any Grade 4 AE Related to IP | 41
  Any Grade 5 AE Related to IP | 2
  Any TEAE Serious Adverse Event (SAE) | 70
  Any SAE Related to IP | 30
  Any TEAE Leading to Stopping of IP | 28
  Any Treatment Related AE Leading to Stopping IP | 16
  Any AE Leading to Dose Reduction | 55
  Any AE Leading to IP Interruption | 81
  Any Treatment Related AE Leading to Dose Reduction | 52
  Treatment Related AE Leading to IP Interruption | 66

ADVERSE EVENTS:
Time Frame: From the first dose of 1enalidomide through 28 days after the last dose of lenalidomide; (maximum duration of study drug was 1940 days).
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 106/134
Serious Adverse Events (participants affected / at risk) | 70/134
Other Adverse Events (participants affected / at risk) | 125/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=134)
ANAEMIA (Blood and lymphatic system disorders) | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 4
ASCITES (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
ENTERITIS (Gastrointestinal disorders) | 1
FAECES DISCOLOURED (Gastrointestinal disorders) | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
PANCREATITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
ASTHENIA (General disorders) | 3
DEATH (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3
MUCOSAL INFLAMMATION (General disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
PYREXIA (General disorders) | 6
SUDDEN DEATH (General disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
ATYPICAL PNEUMONIA (Infections and infestations) | 1
BACTERAEMIA (Infections and infestations) | 2
BACTERIAL SEPSIS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 2
CELLULITIS (Infections and infestations) | 3
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1
H1N1 INFLUENZA (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 8
PNEUMONIA BACTERIAL (Infections and infestations) | 4
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 2
PSEUDOMONAL SEPSIS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 3
SEPTIC SHOCK (Infections and infestations) | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
UROSEPSIS (Infections and infestations) | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 4
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
HEADACHE (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 1
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
URINARY RETENTION (Renal and urinary disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 2
HYPOTENSION (Vascular disorders) | 7
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=134)
ANAEMIA (Blood and lymphatic system disorders) | 42
LEUKOPENIA (Blood and lymphatic system disorders) | 22
LYMPHOPENIA (Blood and lymphatic system disorders) | 10
NEUTROPENIA (Blood and lymphatic system disorders) | 68
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 51
ABDOMINAL PAIN (Gastrointestinal disorders) | 10
CONSTIPATION (Gastrointestinal disorders) | 21
DIARRHOEA (Gastrointestinal disorders) | 45
NAUSEA (Gastrointestinal disorders) | 41
VOMITING (Gastrointestinal disorders) | 16
ASTHENIA (General disorders) | 18
CHILLS (General disorders) | 8
FATIGUE (General disorders) | 47
OEDEMA PERIPHERAL (General disorders) | 22
PYREXIA (General disorders) | 30
NASOPHARYNGITIS (Infections and infestations) | 8
PNEUMONIA (Infections and infestations) | 8
RESPIRATORY TRACT INFECTION (Infections and infestations) | 9
SINUSITIS (Infections and infestations) | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 20
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7
BLOOD CREATININE INCREASED (Investigations) | 7
WEIGHT DECREASED (Investigations) | 20
DECREASED APPETITE (Metabolism and nutrition disorders) | 21
DEHYDRATION (Metabolism and nutrition disorders) | 8
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 19
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
DIZZINESS (Nervous system disorders) | 7
DYSGEUSIA (Nervous system disorders) | 8
HEADACHE (Nervous system disorders) | 8
NEUROPATHY PERIPHERAL (Nervous system disorders) | 9
ANXIETY (Psychiatric disorders) | 11
INSOMNIA (Psychiatric disorders) | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 41
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 24
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8
DRY SKIN (Skin and subcutaneous tissue disorders) | 10
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 23
RASH (Skin and subcutaneous tissue disorders) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Single center publications may not be submitted until after multicenter publication is submitted (or 1 year after study completion), whichever comes first. The investigator may then publish results provided that Celgene receive a copy of any proposed publication/presentation at least 30 days in advance of submission, delete any confidential information & delay the submission for up to 60 additional days for patent filing. Multicenter publications must include input from investigators & Celgene.